CLINICAL TRIAL: NCT05405868
Title: A Phase III, Double-masked, Randomised, Placebo-controlled Trial Investigating the Safety and Efficacy of Nicotinamide (NAM) to Slow Visual Field Loss in Adults With Open-angle Glaucoma
Brief Title: Nicotinamide in Glaucoma (NAMinG): A Randomised, Placebo-controlled, Multi-centre, Phase III Trial
Acronym: NAMinG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTU/2020/365
Record Dates: First submitted 2022-02-25; First posted 2022-06-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma, Open-Angle
Keywords: Nicotinamide; Vitamin B3
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised 1:1 to receive oral Nicotinamide 3g/day or matching Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): Participants will receive Nicotinamide for up to 27 months (treatment period) in addition to an initial treatment of Standard of Care IOP- lowering therapy (prior to randomisation and start of trial treatment) . They will receive 1.5g/day for the first 6 weeks, then dose increase to 3.0g/day for remainder of the treatment period.
  Interventions: Drug: Nicotinomide
- Matching Placebo (Placebo Comparator): Participants will receive matching placebo for up to 27 months (treatment period) in addition to an initial treatment of Standard of Care IOP- lowering therapy (prior to randomisation and start of trial treatment) . They will receive 1.5g/day for the first 6 weeks, then dose increase to 3.0g/day for remainder of the treatment period.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Nicotinomide — Nicotinamide tablets (750mg)
  Arms: Nicotinamide
Drug: Matching placebo — Matching placebo
  Arms: Matching Placebo

SUMMARY:
Glaucoma is the leading cause of sight impairment and blindness worldwide. It is a long-term eye disease which can cause permanent loss of sight and sometimes blindness and affects 1 in 50 people over 50 years of age. Open-angle glaucoma (OAG) is the most common type of glaucoma. This tends to develop slowly over many years, caused by the drainage pathway in the eye gradually becoming blocked over time due to a build-up of fluid. This build-up causes pressure in the eye to increase (intra-ocular pressure (IOP)), which then damages the important nerve at the back of the eye called the optic nerve, resulting in vision loss. Current treatments offered for glaucoma (eye drops or laser surgery), aim to lower eye pressure and have shown to slow vision loss, however, visual disability and blindness rates remain unacceptably high and many patients continue to lose vision despite these treatments, suggesting that the optic nerve in some patients is more easily damaged. Recent research has looked at cells called 'mitochondria'. These cells produce most of the energy in the body, and the nerve cells in the eye need a lot of energy to function and survive. Nicotinamide (NAM) is a form of Vitamin B3 and evidence so far has shown that mitochondrial function can be improved with this treatment. The aim of this trial is to find out whether taking oral NAM when used with current standard treatment for lowering pressure in the eye, can reduce the amount of sight loss in recently diagnosed patients with OAG, and evaluate the long-term safety and effectiveness of NAM. The trial will use two groups of people recently diagnosed with glaucoma and who have normal care (drops or laser) to lower eye pressure. Using a method of randomisation (randomly allocated to each group using a computer system), one group will be given NAM and the other group will be given a placebo or 'dummy pill'. This is a double masked trial meaning the participant nor the Investigator will be told which treatment group patients have been allocated to.

DETAILED DESCRIPTION:
Open Angle Glaucoma (OAG) is a chronic optic neuropathy causing progressive vision loss. It is well established that IOP is the only currently modifiable risk factor for glaucoma progression, and it is widely accepted that other risk factors modulate the susceptibility of an eye to IOP. This has led to a considerable body of research into neurodegenerative mechanisms and potential neuroprotective approaches. Various pathways contributing to the neurodegeneration have been implicated, and many have focussed on the role of mitochondria. Neuroprotection would significantly reduce sight loss and the burden of IOP-lowering eye drop treatment needed for disease control. There is evidence that susceptibility to IOP is related to mitochondrial function and ageing is associated with mitochondrial functional decline. The knowledge gap addressed in this trial is the relative contribution that mitochondrial function makes to glaucomatous neurodegeneration and whether boosting mitochondrial function with NAM slows progression in humans in the same way that it does in animal models. Biomarkers for mitochondrial-related susceptibility have not yet been established in humans. The proposal therefore is a new mechanism neuroprotection to improve resistance to eye pressure and evaluate the long-term safety and efficacy of NAM to preserve vision and its mechanism of action. There is strong evidence that mitochondrial dysfunction is associated with OAG susceptibility and that NAM improves mitochondrial function. Research has shown short-term vision improvement with high-dose NAM in glaucoma patients. NAM is safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been recently diagnosed (within the last 12 months) with early to moderate open-angle glaucoma (OAG) in at least one eye (including primary OAG, normal tension glaucoma (NTG) and pseudoexfoliation glaucoma)
2. Open angle on gonioscopy
3. Adults aged 18 years or over
4. Snellen visual acuity 6/12 or better in at least one eye meeting the visual field (VF) criteria
5. Visual Field (VF) mean deviation (MD) no worse than -12dB in either eye
6. A negative pregnancy test result at the screening and baseline visit prior to randomisation for women of childbearing potential
7. Ability to provide informed consent to participate
8. Able and willing to attend trial visits and comply with trial procedures for the duration of the trial

Exclusion Criteria:

1. Pigment dispersion glaucoma
2. Pregnancy (or planned pregnancy during the trial) and/or breastfeeding
3. Women of childbearing potential and male participants with a partner of childbearing potential not willing to use highly effective contraception for the duration of the trial treatment and for the time period specified following last trial treatment administration.
4. Current treatment with either isoniazid, pyrazinamide, carbamazepine, phenobarbital or primidone
5. Current liver disease or laboratory results with elevated levels of liver transaminases (AST or ALT >3 x ULN) at screening visit.
6. Renal failure (eGFR <30mL/min/1.73m²) at screening visit.
7. Conditions affecting both eyes which may affect the Visual Field test result:

   1. Diabetic retinopathy or any other retinal disease causing VF loss
   2. Clinically relevant cataract (likely to require cataract surgery within the next 2 years)
   3. Dementia or other non-glaucomatous neurological disease causing VF loss
   4. Adnexal conditions causing VF loss (including but not limited to blepharochalasis)
8. Diagnosed with cancer in the last 5 years (with exception of non-melanoma skin cancer).
9. Any clinical condition that, in the investigator's opinion would make the participant unsuitable for the trial.
10. Concurrently enrolled in any other interventional trial or participation in previous clinical trial of glaucoma.
11. Current use of, and unwilling to abstain from, over-the-counter additional vitamin B3/NAM oral supplements (including skin preparations such as ointments/emulsions), Ginkgo Biloba and/or Coenzyme Q10 supplements, throughout the duration of their participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The difference between the treatment arms in change of Visual Field (VF) mean deviation (MD) at 27 months measured by the Humphrey Visual Field Analyser test | Month 27; end of trial treatment
  The Humphrey Visual Field Analyser test is a diagnostic tool commonly used to assess the retina's ability to detect a light stimulus at specific points within the visual field, called retinal sensitivity. Participants will undergo visual field testing at Screening, Baseline, Months 3, 6,12,18, 24 and Month 27 using the Humphrey Visual Field analyser with the SITA Standard 24-2 programme. The results will be used to measure the progression of vision loss between the active arm (Nicotinamide) and the comparator (matching placebo) The primary endpoint will be analysed using a linear mixed model to estimate the difference between treatment groups in VF MD at 27 months. The model will include month 27 VF MD as the outcome and baseline VF MD, IOP-lowering treatment type (eye drops vs laser) and baseline serum NAM levels as covariates.

SECONDARY OUTCOMES:
The difference in Visual Field (VF) mean deviation (MD) at 3 months (0-3 months - neuro-recovery) between the active treatment group and the placebo group, measured using the Humphrey Visual Field analyser test with the SITA Standard 24-2 programme | From Baseline until Month 3
  The Humphrey Visual Field Analyser test is a diagnostic tool commonly used to assess the retina's ability to detect a light stimulus at specific points within the visual field, called retinal sensitivity. Participants will undergo visual field testing using the Humphrey Visual Field analyser with the SITA Standard 24-2 programme. The results will be used to measure the progression of vision loss between the active arm (Nicotinamide) and the comparator (matching placebo) over the initial 0-3 months
Quality-of-Life outcome differences between the two treatment groups at baseline, month 3 and month 27, as measured by the descriptive system for health-related quality of life, EQ-5D-5L with additional vision specific questions. | At Baseline, Month 3 and Month 27
  The EQ-5D-5L (with vision bolt-on) is a participant self-reported questionnaire which evaluates the generic quality of life at the time of completion. It comprises of one question for each of the five dimensions; no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A Visual Analogue Scale is also used and is a scale measured from 0 -100 scale where patients are asked to indicate their overall health on the day of questionnaire completion.
  This version of the questionnaire will also include additional vision related questions as part of the 5 dimensions, known as vision bolt on questions.
Quality-of-Life outcome differences between the two treatment groups at baseline, month 3 and month 27, as measured by the 15-item Glaucoma Quality of Life Questionnaire. | At Baseline, Month 3 and Month 27
  The Glaucoma Quality of Life Questionnaire (GQL-15) is a 15-item which measures the severity of visual disability and comprises of 15 vision-related items. The item-level responses for each factor are coded on a five-point scale (1 meaning no difficulty and 5 meaning severe difficulty), while 0 is marked if the participant does not perform the activity as a result of non-visual cause. These items are grouped into four subscales: 1) "Central and near vision" (two items); 2) "Peripheral vision" (six items); 3) "Dark adaptation and glare" (six items); and 4) "Outdoor mobility" (one item). Total score is derived by summing all item-level response scores.
The safety profile of high dose NAM, measured by liver function tests (LFTs) at Screening, Month 3 and Month 18 | At Screening, Month 3 and Month 18
  The Liver Function test is a standard diagnostic laboratory assay used to diagnose and monitor liver disease or damage. The tests measure the levels of certain enzymes and proteins in the blood.
The safety profile of high dose NAM, measured from blood glucose test, HbA1c at Screening, Month 3 and Month 18 | At Screening, Month 3 and Month 18
  The HbA1c blood test is a standard diagnostic laboratory test used to measure blood sugar levels.
The safety profile of high dose NAM, measured by estimated glomerular filtration rate (eGFR) at Screening, Month 3 and Month 18 | At Screening, Month 3 and Month 18
  The eGFR blood test is a standard diagnostic laboratory test used to measure how well the kidney function is.
The number of adverse events as assessed by CTCAE v5.0 from baseline to month 27 | From Baseline until end of trial treatment and trial completion at Month 27
  Number of participants with treatment related adverse events assessed by CTCAE v5.0 from baseline to month 27.

OTHER OUTCOMES:
The impact of NAM treatment on mitochondrial function in the active treatment group between baseline and month 27, measured using the Seahorse mitochondrial function test. | From Baseline until end of trial treatment at Month 27
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples. NAM, which is a form of Vitamin B3 is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells.
The impact of NAM treatment on mitochondrial function in the placebo group between baseline and month 27, measured using the Seahorse mitochondrial function test. | From Baseline until end of trial treatment at Month 27
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples. NAM, which is a form of Vitamin B3 is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells.
The association between lymphocyte mitochondrial function, measured by the Seahorse mitochondrial function test, and rate of visual field loss in the placebo group between baseline and month 27. | From Baseline until end of trial treatment at Month 27
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples. Mitochondrial function will be regarded as time-varying covariate and a repeated measures model will be used.
The association between nicotinamide adenine dinucleotide levels, from peripheral blood mononuclear cells, and the rate of visual field loss in the placebo group between baseline and month 27. | From Baseline until end of trial treatment at Month 27
  Nicotinamide (NAM) is a major precursor of nicotinamide adenine dinucleotide (NAD) in neurones. NAD is an essential cofactor in oxidative phosphorylation and adenosine triphosphate (ATP) production. It plays a central role in mitochondrial function.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure NAD. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque). Mitochondrial function will be regarded as time-varying covariate and a repeated measures model will be used.
Test the hypothesis that lower mitochondrial function, measured using the Seahorse mitochondrial function test, is associated with lower nicotinamide (NAM) levels collected from vitamin B3 blood samples in the placebo group at baseline | Baseline only
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples. NAM levels is the measure of Vitamin B3, which is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
Test the hypothesis that lower mitochondrial function, measured using the Seahorse mitochondrial function test, is associated with lower nicotinamide (NAM) levels collected from vitamin B3 blood samples in the active treatment group at baseline | Baseline only
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples. NAM levels is the measure of Vitamin B3, which is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
Test hypothesis that lower mitochondrial function, measured by the Seahorse mitochondrial function test, is associated with lower nicotinamide adenine dinucleotide levels collected from peripheral blood mononuclear cells in the placebo group at baseline | Baseline only
  Nicotinamide (NAM) is a major precursor of nicotinamide adenine dinucleotide (NAD) in neurones. NAD is an essential cofactor in oxidative phosphorylation and adenosine triphosphate (ATP) production. It plays a central role in mitochondrial function. Low levels of NAD are associated with low levels of mitochondrial function.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure NAD. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
Test hypothesis that lower mitochondrial function, measured by the Seahorse mitochondrial function test, is associated with lower nicotinamide adenine dinucleotide levels collected from PBMC blood samples in the active treatment group at baseline | Baseline only
  Nicotinamide (NAM) is a major precursor of nicotinamide adenine dinucleotide (NAD) in neurones. NAD is an essential cofactor in oxidative phosphorylation and adenosine triphosphate (ATP) production. It plays a central role in mitochondrial function. Low levels of NAD are associated with low levels of mitochondrial function.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure NAD. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
Test the hypothesis that lower mitochondrial function, measured using the Seahorse mitochondrial function test, is associated with higher oxidised glutathione levels collected from peripheral blood mononuclear cells in the placebo group at baseline | Baseline only
  Glutathione is an antioxidant produced in cells and any imbalance can cause oxidative stress. High oxidative stress levels can be a precursor to disease and it is associated with lower mitochondrial function.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure glutathione. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
Test hypothesis that lower mitochondrial function, measured using the Seahorse mitochondrial function test, is associated with higher oxidised glutathione levels collected from PBMC blood samples in the active treatment group at baseline | Baseline only
  Glutathione is an antioxidant produced in cells and any imbalance can cause oxidative stress. High oxidative stress levels can be a precursor to disease and it is associated with lower mitochondrial function.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure glutathione. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
The connection between nicotinamide (NAM) levels, measured from vitamin B3 blood samples, and the EPIC Food Frequency Questionnaire responses in the placebo group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  NAM levels is the measure of Vitamin B3, which is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
The connection between nicotinamide (NAM) levels, measured from vitamin B3 blood samples, and the EPIC Food Frequency Questionnaire responses in the active treatment group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  NAM levels is the measure of Vitamin B3, which is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
The connection between NAD levels, measured from peripheral blood mononuclear cells, and the EPIC Food Frequency Questionnaire responses in the placebo group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure NAD. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
The connection between NAD levels, measured from peripheral blood mononuclear cells, and the EPIC Food Frequency Questionnaire responses in the active treatment group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure NAD. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
The connection between oxygen consumption rate (OCR) levels, measured from peripheral blood mononuclear cells, and the EPIC Food Frequency Questionnaire responses in the placebo group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure OCR. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
The connection between oxygen consumption rate (OCR) levels, measured from peripheral blood mononuclear cells, and the EPIC Food Frequency Questionnaire responses in the active treatment group at baseline | Baseline only
  The EPIC Food Frequency Questionnaire (FFQ) is to measure a participant's usual food intake during the previous year and will help identify the intake level and absorption of Vitamin B3 via natural sources of food.
  Peripheral blood mononuclear cell (PBMC) are used to measure immunological functions and will be used to measure OCR. Cells are isolated from blood samples using standardised density gradient technique (Ficoll-Paque).
The effect of NAM on the rate of visual field loss between Month 3 and Month 27,measured by the Humphrey Visual Field Analyser test | From Month 3 until end of trial treatment at Month 27
  The Humphrey Visual Field Analyser test is a diagnostic tool commonly used to assess the retina's ability to detect a light stimulus at specific points within the visual field, called retinal sensitivity.
The effect of NAM on the level of mitochondrial function in participants with low vs high baseline mitochondrial function and low vs high baseline NAM levels between month 3 and month 27, measured from Vitamin B3 blood samples . | From Baseline until end of trial treatment at Month 27
  The Vitamin B3 is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
The association between lymphocyte mitochondrial function, measured by the Seahorse mitochondrial function test, and quality of life measures, as measured by the EQ-5D-5L and GQL-15 questionnaires, in the placebo group between baseline and month 27. | From Baseline until end of trial treatment at Month 27
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples.
The association between lymphocyte mitochondrial function, measured by the Seahorse mitochondrial function test, and quality of life measures, measured by the EQ-5D-5L and GQL-15, in the active treatment group between baseline and month 27. | From Baseline until end of trial treatment at Month 27
  The Seahorse mitochondrial function test measures oxygen during energy production processes that occur in the mitochondria by directly measuring the oxygen consumption rate (OCR) of cells. The measurement will be performed on Peripheral Blood Mononuclear Cell (PBMC) blood samples.
The association between baseline NAM levels and rate of visual field loss in the placebo group between baseline and month 27, as measured by the Humphrey Visual Field Analyser test and Vitamin B3 blood samples. | From Baseline until end of trial treatment at Month 27
  The Humphrey Visual Field Analyser test is a diagnostic tool commonly used to assess the retina's ability to detect a light stimulus at specific points within the visual field, called retinal sensitivity.
  The Vitamin B3 is crucial for cell metabolism, normal functioning of the central nervous system and the formation of red blood cells. The vitamin B3 blood test is a standard diagnostic laboratory test used to measures the level of vitamin B3 in the blood and to determine Vitamin B3 (Niacin) deficiencies.
The association between NAM dosing and IOP in the active and placebo groups between baseline and month 27, measured by applanation tonometers . | From Baseline until end of trial treatment Month 27
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method used to determine the fluid pressure inside the eye (Intraocular pressure (IOP)) in the evaluation of patients at risk of glaucoma. Most tonometers are calibrated to measure pressure in millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: David Garway-Heath, Principal Investigator — UCL
Locations (10):
- United Kingdom (10):
  - Belfast City Hospital, Belfast, Northern Ireland
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Queen Victoria Hospital NHS Foundation Trust, East Grinstead
  - Royal Liverpool Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Barnet Hospital, Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Manchester Royal Eye Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD has been made at this time